CLINICAL TRIAL: NCT04905550
Title: An Exploratory Clinical Study of Almonertinib in Combination With Craniocerebral Radiotherapy in First-line Treatment of EGFR Positive Non-Small Cell Lung Cancer(NSCLC) With Brain Metastases
Brief Title: Almonertinib Combined With Cerebral Radiation Treat Brain Metastases From EGFR Positive NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ying Wang, Associate Director of Chongqing University Cancer Hospital, Chongqing University Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RadiAl-CNS
Record Dates: First submitted 2021-05-23; First posted 2021-05-27 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
Keywords: Almonertinib; Radiotherapy; Brain Metastasis; Non-Small Cell Lung Cancer; Intracranial Progress Free Survival
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — aumolertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Craniocerebral radiotherapy combined with Almonertinib 110mg p.o qd (Experimental): Almonertinib mesylate tablet, 110mg, qd; until the disease progresses or unacceptable toxicity.
  The craniocerebral radiotherapy was acceptable from 1 week before to 6 weeks after treatment with Almonertinib.
  Dose adjustment and delay of Almonertinib are allowed. Delay of Almonertinib is allowed for up to 9 weeks, calculated from the time of last administration, otherwise, treatment is terminated.
  Interventions: Drug: Almonertinib; Radiation: Stereotactic Radiotherapy(SRT) or Stereotactic Radiosurgery(SRS) or Whole-Brain Radiotherapy(WBRT)

INTERVENTIONS:
Drug: Almonertinib — Almonertinib 110mg p.o qd. Treatment with Almonertinib will continue until progression or unacceptable toxicity.
  Other Names: The third generation of EGFR - TKI
Radiation: Stereotactic Radiotherapy(SRT) or Stereotactic Radiosurgery(SRS) or Whole-Brain Radiotherapy(WBRT) — Image guided, 24-15 Gy*1F was recommended if use SRS. 9-12 Gy*3F/1W or 6Gy×5F/1W was recommended if use SRT. 30Gy/10F/2W for WBRT, large residual lesions will be treated with a local dose (≤DT 45Gy/15F).

SUMMARY:
According to literature reports, about 16.3%-19% of newly diagnosed NSCLC patients are associated with brain metastasis, and 30%-50% of NSCLC patients will develop brain metastasis during the whole course of the disease.

Patients with EGFR positive-type had a 10-15% higher risk of brain metastasis than patients with EGFR wild-type. mOS in patients with EGFR positive were twice as high as those with EGFR wild-type, despite the presence of brain metastasis.

Improving the control rate of intracranial lesions in patients with EGFR positive can not only improve the quality of life, but also may translate into survival benefits and improve OS. Previous studies have shown that in lung cancer patients with EGFR-sensitive mutations, craniocerebral radiotherapy prior to delayed craniocerebral radiotherapy significantly prolonged OS.

The first-line treatment of the third generation of EGFR-TKI targeting drug Almonertinib for EGFR-positive NSCLC can eliminate the possible EGFR T790M mutant clones at an early stage and better control the disease progression. Moreover, Almonertinib is easy to pass through the blood-brain barrier, which can not only better control intracranial lesions, but also control, prevent or delay the occurrence of brain metastasis.

This study was intended to conduct a randomized controlled study on the safety and efficacy of early craniocerebral radiotherapy combined with Almonertinib in patients with EGFR positive non-small cell lung cancer with brain metastasis.

Through the above studies we hope to confirm that early craniocerebral radiotherapy combined with Almonertinib is safe and feasible for patients with EGFR positive newly diagnosed with brain metastasis, and can prolong the intracranial progression-free survival (IPFS), and even extend the progression-free survival (PFS) and overall survival (OS).

DETAILED DESCRIPTION:
All eligible patients will receive craniocerebral radiotherapy in combination with Almonertinib.

Here are two types of craniocerebral radiotherapy:

1. SRS or SRT is recommended for patients with ≤4 intracranial metastases and the maximum lesion ≤4cm. 24-15 Gy*1F was recommended if use SRS. 9-12 Gy*3F or 6Gy×5F was recommended if use SRT.
2. For >4 intracranial metastases, or the maximum lesion>4cm, whole-brain radiotherapy (WBRT) of 30Gy/10F was recommended, and then the large residual lesions will be treated with a local dose (≤DT 45Gy/15F). Hippocampal protection is highly recommended.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old (calculated from the time when the subject signed the informed consent), both male and female.
2. Confirmed pathology of EGFR mutation positive（exon 19 deletion, L858R, T790M）NSCLC with brain metastases on enhanced MRI.
3. Subjects had not previously received chemotherapy, EGFR-TKI, biologic or immunotherapy, or other experimental therapy as first-line treatment for advanced NSCLC.
4. According to RECIST 1.1 criteria, subjects must have a measurable target lesion (maximum diameter under MRI/CT ≥10mm, short diameter of lymph node ≥15mm) that has been examined by CT or MRI.Tumor imaging evaluation was performed within 28 days prior to initial treatment.
5. ECOG PS score: 0-1 points.
6. Must be able to swallow tablets，and expected survival ≥3 months.
7. Clinical diagnosis of Alzheimer's patients who can be treated with radiation therapy.
8. All screening laboratory tests are performed according to protocol and need to be performed within 14 days prior to the first dose.The values of laboratory tests performed by screening must meet the following criteria:

   1. Routine blood examination :(no blood transfusion, no G-CSF, no drug correction within 14 days before screening)

      * Hemoglobin (Hb) ≥90 g/L;
      * Absolute neutrophil count (ANC) ≥1.5×109/L;
      * Platelet count (PLT) ≥100×109/L;
      * White blood cell count (WBC) ≥4.0×109/L and ≤15×109/L;
   2. Biochemical test :(no blood transfusion or albumin within 14 days prior to screening)

      * AST and ALT ≤1.5×ULN (such as cancer that has spread to the liver, ≤5×ULN);
      * ALP≤2.5×ULN (such as tumor bone metastases, ≤5×ULN);
      * TBiL≤1.5×ULN.
      * ALB≥30 g/L;
      * Cr≤1.5×ULN, while creatinine clearance (CrCL)≥60 mL/min (Cockcroft - Gault formula);
      * APTT≤1.5×ULN, at the same time of INR or PT≤1.5×ULN (without anticoagulation therapy).
9. Women of childbearing age must have a serum pregnancy test within 3 days prior to the first dose and the results are negative.Women of reproductive age subjects and male subjects whose partners are women of reproductive age must agree to use barrier contraception (i.e., condoms) during the study period and for 180 days after the last administration of the study drug.
10. Volunteered to participate in clinical studies and signed informed consent.

Exclusion Criteria:

1. Exclusion criteria for target diseases:

   1. Subjects who had previously received anti-EGFR-TKI therapy.
   2. Patients with neuromeningeal disease but no intracranial metastases confirmed by MRI and/or CSF malignancy.
   3. Previous radiotherapy for CNS metastases, including measurable or unmeasurable sites of the disease for efficacy assessment.
   4. Patients who had undergone a major surgical procedure (other than placement of vascular access or CNS shunt) or had a major traumatic injury or were expected to require major surgery during the study period within 4 weeks prior to initial dosing.
   5. Subject who can be surgically excised or treated with radical radiotherapy.
2. History and complications:

   1. The patient is using (or cannot be discontinued for at least 1 week prior to the first dosing of the investigational treatment) some drug or herbal supplement known to be a strong depressant or inducer of CYP3A4/5 (Appendix 8).
   2. Excluding uncontrollable nausea and vomiting, chronic gastrointestinal disease, prior gastrectomy or other surgery, may affect the full absorption of the study drug.
   3. exclude the presence of any serious or uncontrolled systemic disease or condition, including:

      * Uncontrolled high blood pressure, diabetes, thyroid disease;
      * Severe heart, lung or kidney disease;
      * Active bleeding constitution;
      * Any bacterial, viral, fungal or other active infection that the Investigator considers to pose a serious risk to the patient;
      * Active hepatitis (HBsAg positive or HBcAb positive, HBV DNA positive), or HCV antibody positive or HIV positive.
   4. Patients with unstable symptomatic metastases: Any unstable and symptomatic CNS or distant metastases that were not controlled by previous surgery, radiotherapy, or corticosteroid treatment within 2 weeks prior to the initial study treatment.Corticosteroids were used before treatment for CNS symptoms, but the symptoms were controllable after treatment, and corticosteroids were used during radiotherapy.
   5. Exclude subjects who are participating in other clinical studies or whose first administration has been less than 3 weeks (or 5 half-lives of the investigational drug) since the end of the previous clinical study (last dosing).
   6. Excluding subjects who expected to require any other form of antitumor therapy (including maintenance therapy with other NSCLC drugs, and/or surgical resection) during the study.
   7. excluded subjects with high suspicion of interstitial pneumonia; Or subjects that may interfere with the detection or management of suspected drug-related pulmonary toxicity;Or other moderate to severe lung diseases that seriously affect lung function.
   8. Subjects with other active malignancies requiring concurrent treatment were excluded.
   9. Subjects with a previous history of malignancy were excluded unless they had achieved a complete response at least 5 years prior to screening and did not require or are not expected to require additional treatment during the study period for basal cell carcinoma of the skin, superficial bladder carcinoma, squamous cell carcinoma of the skin, or cervical carcinoma in situ.Rule out with Ⅱ magnitude myocardial ischemia and myocardial infarction, arrhythmia of the subjects of poor control.
   10. Ruled out according to the NYHA standard Ⅲ ~ Ⅳ level cardiac insufficiency or heart colour to exceed examination: LVEF, left ventricular ejection fraction < 50% of the subjects.
   11. Patients with significant hemoptysis or hemoptysis of half a teaspoon (2.5ml) or more per day within 1 month before randomization.
   12. Patients with bleeding symptoms of significant clinical significance or with definite bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, or vasculitis, occurred within 1 month prior to randomization.
   13. Artery/venous thrombosis events occurred in the first 3 months at random, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism, etc.
   14. Subjects with active tuberculosis (TB) were excluded.In subjects suspected of active TB, chest X-rays and sputum should be examined, and clinical signs and symptoms should be excluded.Subjects with a history of active tuberculosis infection within the previous 1 year were screened, even if they had been treated. Subjects with a history of active TB infection more than 1 year ago should also be excluded unless the course and type of anti-TB treatment previously used is demonstrated to be appropriate.
   15. Excluding subjects who were preparing for or had previously received tissue/organ transplants.
   16. Subjects who received or will receive live vaccine within 30 days prior to the first dose were excluded.
   17. Inclusion of subjects with uncontrolled tumor-related pain is not recommended.Subjects requiring pain medication must have a stable pain control regimen;Symptomatic lesions suitable for palliative radiotherapy (such as bone metastases or nerve invasion metastases) should be completed at least 2 weeks before inclusion; Asymptomatic metastatic foci whose further growth may result in dysfunction or intractable pain (e.g. epidural metastases that do not show spinal cord compression) should be considered for local-regional treatment before randomization, if appropriate.
3. Physical examination and laboratory examination

   1. A known history of positive human immunodeficiency virus (HIV) tests or a known history of acquired immunodeficiency syndrome (AIDS).
   2. Untreated active hepatitis:

      * Hepatitis B: HBV surface antigen (HBV sAg) positive and HBV DNA detection value is higher than the upper limit of normal value;
      * Hepatitis C: Hepatitis C virus antibody (HCV Ab) positive, HCV RNA positive, and abnormal liver function;
      * Complicated with hepatitis B and C co-infection.
   3. Exclude subjects with uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
4. Allergic reactions and adverse drug reactions:Study drugs with CYP3A4 inhibition agents, inducers, or drugs with a narrow therapeutic window that are CYP3A4-sensitive substrates were used within 7 days before the first administration.
5. Patients receiving concurrent chemotherapy were excluded.
6. Excludes subjects with mental illness, alcoholism, inability to quit smoking, drug or substance abuse.
7. At the discretion of the Investigator, exclude subjects with history or current evidence of any disease, treatment or laboratory anomaly that may confuse study results, interfere with subjects' participation in the study procedure, or is not in the best interest of subjects' participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Intracranial Progress Free Survival(iPFS) | Up to 4 years
  As determined by the investigator using RECIST 1.1 criteria between patients receiving Almonertinib and craniocerebral radiotherapy. iPFS is defined as The time between the start of treatment and the observation of progression of intracranial lesions or death from any cause. In order to ascertain this endpoint, efforts will be made so that patients will be followed for 156 weeks or until progression of disease (and treatment cessation), whichever comes first. At each time-point, subjects should have CT/MR of chest and head with contrast.

SECONDARY OUTCOMES:
Number of adverse events of grade 3-4 or higher | Up to 4 years
  To estimate and compare rates of ≥ grade 3-4 adverse events, by organ system, by CTCAEv4.0 that occur within 3 months from the start of craniocerebral radiotherapy when given prior to or concurrently with Almonertinib.
Rate of long term adverse events | Up to 4 years
  To estimate and compare the rates of long-term adverse events (after 3 months) from the end of craniocerebral radiotherapy when given prior to or concurrently with Almonertinib.
Rate of change in tumor microenvironment | Up to 4 years
  To evaluate and compare changes in the tumor microenvironment induced by radiation when given prior to or concurrently with Almonertinib.
Changes in EGFR mutations | Up to 4 years
  To evaluate whether response to therapy correlates with changes in EGFR mutations among patients treated with Almonertinib combined with craniocerebral radiotherapy.
Overall Survival | Up to 4 years
  Time from entry to death from any cause (the last follow-up time for patients lost to follow-up; Patients who were still alive at the end of the study, the end date of follow-up).

CONTACTS AND LOCATIONS:
Overall Officials: Ying Wang, Ph.D, M.D., Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagasaka M, Zhu VW, Lim SM, Greco M, Wu F, Ou SI. Beyond Osimertinib: The Development of Third-Generation EGFR Tyrosine Kinase Inhibitors For Advanced EGFR+ NSCLC. J Thorac Oncol. 2021 May;16(5):740-763. doi: 10.1016/j.jtho.2020.11.028. Epub 2020 Dec 15. PMID 33338652
- [Background] Dong RF, Zhu ML, Liu MM, Xu YT, Yuan LL, Bian J, Xia YZ, Kong LY. EGFR mutation mediates resistance to EGFR tyrosine kinase inhibitors in NSCLC: From molecular mechanisms to clinical research. Pharmacol Res. 2021 May;167:105583. doi: 10.1016/j.phrs.2021.105583. Epub 2021 Mar 26. PMID 33775864
- [Background] Wakuda K, Yamaguchi H, Kenmotsu H, Fukuda M, Takeshita M, Suetsugu T, Kirita K, Ebi N, Hataji O, Miura S, Chibana K, Okamoto I, Yoshimura K, Nakagawa K, Yamamoto N, Sugio K. A phase II study of Osimertinib for patients with radiotherapy-naive CNS metastasis of non-small cell lung cancer: treatment rationale and protocol design of the OCEAN study (LOGIK 1603/WJOG 9116L). BMC Cancer. 2020 May 1;20(1):370. doi: 10.1186/s12885-020-06874-6. PMID 32357848
- [Background] Franchino F, Ruda R, Soffietti R. Mechanisms and Therapy for Cancer Metastasis to the Brain. Front Oncol. 2018 May 24;8:161. doi: 10.3389/fonc.2018.00161. eCollection 2018. PMID 29881714
- [Background] Nishino M, Soejima K, Mitsudomi T. Brain metastases in oncogene-driven non-small cell lung cancer. Transl Lung Cancer Res. 2019 Nov;8(Suppl 3):S298-S307. doi: 10.21037/tlcr.2019.05.15. PMID 31857953
- [Background] Nieder C, Norum J, Dalhaug A, Aandahl G, Pawinski A. Radiotherapy versus best supportive care in patients with brain metastases and adverse prognostic factors. Clin Exp Metastasis. 2013 Aug;30(6):723-9. doi: 10.1007/s10585-013-9573-x. Epub 2013 Feb 8. PMID 23392634
- [Background] Andrews DW, Scott CB, Sperduto PW, Flanders AE, Gaspar LE, Schell MC, Werner-Wasik M, Demas W, Ryu J, Bahary JP, Souhami L, Rotman M, Mehta MP, Curran WJ Jr. Whole brain radiation therapy with or without stereotactic radiosurgery boost for patients with one to three brain metastases: phase III results of the RTOG 9508 randomised trial. Lancet. 2004 May 22;363(9422):1665-72. doi: 10.1016/S0140-6736(04)16250-8. PMID 15158627
- [Background] Chang JY, Bezjak A, Mornex F; IASLC Advanced Radiation Technology Committee. Stereotactic ablative radiotherapy for centrally located early stage non-small-cell lung cancer: what we have learned. J Thorac Oncol. 2015 Apr;10(4):577-85. doi: 10.1097/JTO.0000000000000453. PMID 25514807
- [Background] Gomez DR, Blumenschein GR Jr, Lee JJ, Hernandez M, Ye R, Camidge DR, Doebele RC, Skoulidis F, Gaspar LE, Gibbons DL, Karam JA, Kavanagh BD, Tang C, Komaki R, Louie AV, Palma DA, Tsao AS, Sepesi B, William WN, Zhang J, Shi Q, Wang XS, Swisher SG, Heymach JV. Local consolidative therapy versus maintenance therapy or observation for patients with oligometastatic non-small-cell lung cancer without progression after first-line systemic therapy: a multicentre, randomised, controlled, phase 2 study. Lancet Oncol. 2016 Dec;17(12):1672-1682. doi: 10.1016/S1470-2045(16)30532-0. Epub 2016 Oct 24. PMID 27789196
- [Background] Garon EB, Siegfried JM, Stabile LP, Young PA, Marquez-Garban DC, Park DJ, Patel R, Hu EH, Sadeghi S, Parikh RJ, Reckamp KL, Adams B, Elashoff RM, Elashoff D, Grogan T, Wang HJ, Dacic S, Brennan M, Valdes Y, Davenport S, Dubinett SM, Press MF, Slamon DJ, Pietras RJ. Randomized phase II study of fulvestrant and erlotinib compared with erlotinib alone in patients with advanced or metastatic non-small cell lung cancer. Lung Cancer. 2018 Sep;123:91-98. doi: 10.1016/j.lungcan.2018.06.013. Epub 2018 Jun 22. PMID 30089602
- [Result] Yang JC, Camidge DR, Yang CT, Zhou J, Guo R, Chiu CH, Chang GC, Shiah HS, Chen Y, Wang CC, Berz D, Su WC, Yang N, Wang Z, Fang J, Chen J, Nikolinakos P, Lu Y, Pan H, Maniam A, Bazhenova L, Shirai K, Jahanzeb M, Willis M, Masood N, Chowhan N, Hsia TC, Jian H, Lu S. Safety, Efficacy, and Pharmacokinetics of Almonertinib (HS-10296) in Pretreated Patients With EGFR-Mutated Advanced NSCLC: A Multicenter, Open-label, Phase 1 Trial. J Thorac Oncol. 2020 Dec;15(12):1907-1918. doi: 10.1016/j.jtho.2020.09.001. Epub 2020 Sep 9. PMID 32916310